CLINICAL TRIAL: NCT05005221
Title: Single Center, Pilot Evaluation of Home-based Therapeutic Drug Monitoring for Tacrolimus and Mycophenolate in Kidney Transplantation
Brief Title: Home-based Therapeutic Drug Monitoring in Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Manjunath Prakash Pai, Professor of Clinical Pharmacy, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00198148
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Kidney Transplant
Keywords: Tacrolimus; Mycophenolate; Therapeutic Drug Monitoring

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:2 allocation ratio to receive one of two text messaging interventions (basic text message reminders or more intensive bidirectional messages).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unidirectional Text Reminders (Active Comparator): Participants in the unidirectional text reminder arm will receive automated text messages to remind them to collect blood samples 48 hours before, 12 hours before, and the morning of the planned sample collection.
  N=15
  Interventions: Behavioral: Automated text messages
- Bidirectional Text Communication (Experimental): Participants in the bidirectional text communication arm will also receive automated messages to remind them to collect blood samples 48 hours before, 12 hours before, and the morning of the planned sample collection but they will be asked to confirm the planned day or reschedule. On the day of sample collection participants will also reply with the time the samples are collected to trigger future reminder messages for each of the 4 samples.
  N=30
  Interventions: Behavioral: Automated text messages

INTERVENTIONS:
Behavioral: Automated text messages — Automated text messages will be used to facilitate blood sample collection at home for therapeutic drug monitoring of tacrolimus and mycophenolate. Participants will collect dried blood samples on 4 occasions. Two days in the clinical with simultaneous venipuncture (one sample) and two days at home with 4 samples collected at specified time points over 8 hours.

SUMMARY:
This is a randomized clinical trial to assess an intervention to facilitate patient self-collection of dried blood samples at home for therapeutic drug monitoring of tacrolimus and mycophenolate in kidney transplant recipients.

In this study, text messages will be sent to mobile devices to remind kidney transplant recipients to perform therapeutic drug monitoring at home using a special lancet device to collect blood samples from the upper arm. The primary objective is to evaluate if more intensive, bidirectional text messages improve the quality of sample collection.

DETAILED DESCRIPTION:
Optimal immunosuppression therapy, most commonly with tacrolimus and mycophenolate, is critical for kidney transplantation success. While graft and patient survival are multifaceted phenomena, they are commonly attributed to chronic, subclinical immune-mediated damage, tacrolimus nephrotoxicity, or premature death secondary to complications amplified by immunosuppression such as infection, malignancy, and cardiovascular disease. New approaches are required to explore ways to optimize the precision dosing of immunosuppression to reduce the associated significant long-term side effects with the potential to improve kidney transplantation outcomes.

Currently, immunosuppressant dose adjustments empirically balance efficacy and toxicity in conjunction with limited tacrolimus blood concentrations. However, both tacrolimus and mycophenolate possess interpatient variability in drug exposure and response with considerable overlap between therapeutic and adverse effects. Only tacrolimus is routinely monitored as mycophenolate trough concentration is not correlated with drug exposure or outcomes. The pharmacokinetic parameter area under the concentration-time curve (AUC) offers a greater understanding of total drug exposure and has been associated with improved outcomes for both tacrolimus and mycophenolate. Yet, AUC is not routinely determined because it is impractical due to the need for multiple repeated samples in the clinic.

The investigators propose a prospective, single-center pilot study to evaluate the ability of a text messaging intervention coupled with a novel lancet device, the Tasso-M20, to facilitate the collection of dried blood samples by the patient at home for AUC estimation. The goal of the project is to develop a patient-centric strategy to allow frequent, longitudinal, minimally invasive sample collection which allows for more detailed assessments of immunosuppression exposure.

The primary objective is to compare the effect of bidirectional text communication on adherence to and accuracy of home-based AUC collection versus unidirectional text reminders in kidney transplant recipients receiving tacrolimus and mycophenolate.

The secondary objective is to assess the bioanalytical agreement of two sample collection methods (dried blood spot and venipuncture) as measured by Liquid Chromatography with tandem mass spectrometry (LC-MS/MS).

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a kidney or kidney/pancreas transplant
* Receiving immediate-release tacrolimus and mycophenolate mofetil
* Willing to received text messages with a mobile device capable of receiving messages
* Willing to receive standard labs at a Michigan Medicine lab draw site on 2 occasions
* Ability to understand, read, and speak English
* Ability to understand and willingness to sign written informed consent

Exclusion Criteria:

* History of multi-organ transplant (other than pancreas)
* History of allergy to tape adhesives

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Unidirectional Text Reminders: Participants in the unidirectional text reminder arm received automated text messages to remind them to collect blood samples 48 hours before, 12 hours before, and the morning of the planned sample collection.
- Bidirectional Text Communication: Participants in the bidirectional text communication arm received automated messages to remind them to collect blood samples 48 hours before, 12 hours before, and the morning of the planned sample collection but they were asked to confirm the planned day or reschedule. On the day of sample collection participants also replied with the time the samples are collected to trigger future reminder messages for each of the 4 samples.
- Analytical Validation: Participants in analytical validation group provided paired dried and venous blood.
Period: Overall Study
Arm/Group | Unidirectional Text Reminders | Bidirectional Text Communication | Analytical Validation
Started | 5 | 9 | 27
Completed | 5 | 9 | 25
Not Completed | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unidirectional Text Reminders | Bidirectional Text Communication | Analytical Validation | Total
Number analyzed (Participants) | 5 | 9 | 25 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (10.2) | 52.3 (8.8) | 54 (14.4) | 53.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6 | 12
  Male | 3 | 5 | 19 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 9 | 25 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percent of Samples Successfully Returned for Drug Monitoring by Participants in the Unidirectional and Bidirectional Arms
Description: Successful home-based therapeutic drug monitoring is defined as a binary composite of 1) timely receipt (postmarked within 48 hours of planned sample collection) of samples and 2) adequate documentation of sample collection time data for pharmacokinetic analysis. Each participant in the Unidirectional and Bidirectional Text Communication arms had two opportunities for sample collection. Participants in the third arm for bioanalytical validation did not complete home sample collection and do not have results for this outcome measure.
Time Frame: 3 months
Population: Participants in Unidirectional and Bidirectional text communication arms
Measure: Number; unit: % of samples postmarked with 48 hrs
Units Other Than Participants: samples
Groups:
- Unidirectional Text Reminders: Participants in the unidirectional text reminder arm will receive automated text messages to remind them to collect blood samples 48 hours before, 12 hours before, and the morning of the planned sample collection.
- Bidirectional Text Communication: Participants in the bidirectional text communication arm will also receive automated messages to remind them to collect blood samples 48 hours before, 12 hours before, and the morning of the planned sample collection but they will be asked to confirm the planned day or reschedule. On the day of sample collection participants will also reply with the time the samples are collected to trigger future reminder messages for each of the 4 samples.
Arm/Group | Unidirectional Text Reminders | Bidirectional Text Communication
Number analyzed (Participants) | 5 | 9
Number analyzed (samples) | 10 | 18
% of samples postmarked with 48 hrs | 83 | 100

2. Secondary Outcome: Percent of Paired Samples With </=15% Difference Between Tacrolimus Concentrations Obtained Via Dried Blood and Venipuncture in the Analytical Validation Arm
Description: Compare concentrations of tacrolimus obtained using the two sample collection methods (dried blood and venipuncture) as measured by liquid chromatography with tandem mass spectrometry (LC-MS/MS). Each participant in the analytical validation arm provided two sets of paired samples on different days.
Time Frame: 2 days
Population: Participants from the analytical validation arm
Measure: Number; unit: % of pairs with %difference </=15%
Units Other Than Participants: sample pairs
Groups:
- Analytical Validation: Participants in analytical validation group provided paired dried and venous blood. Each participant provided 2 samples on different days.
Arm/Group | Analytical Validation
Number analyzed (Participants) | 25
Number analyzed (sample pairs) | 50
% of pairs with %difference </=15% | 80

3. Secondary Outcome: Percent of Paired Samples With </=15% Difference Between Mycophenolic Acid Concentrations Obtained Via Dried Blood and Venipuncture in the Analytical Validation Arm
Description: Compare concentrations of mycophenolic acid obtained using the two sample collection methods (dried blood and venipuncture) as measured by liquid chromatography with tandem mass spectrometry (LC-MS/MS). Each participant in the analytical validation arm provided two sets of paired samples on different days.
Time Frame: 2 days
Population: Participants from the analytical validation arm
Measure: Number; unit: % of pairs with %difference </=15%
Units Other Than Participants: sample pairs
Arm/Group | Analytical Validation
Number analyzed (Participants) | 25
Number analyzed (sample pairs) | 50
% of pairs with %difference </=15% | 76

ADVERSE EVENTS:
Time Frame: 48 hours after sample collection
Arm/Group | Unidirectional Text Reminders | Bidirectional Text Communication | Analytical Validation
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/9 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/9 | 0/25
Other Adverse Events (participants affected / at risk) | 0/5 | 0/9 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT05005221/Prot_SAP_000.pdf